CLINICAL TRIAL: NCT02319304
Title: Phase II Trial of Low Dose Whole Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX for Patients With Newly Diagnosed T3N0M0, T2N1M0, or T3N1M0 Rectal Adenocarcinoma
Brief Title: Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX for Patients With Newly Diagnosed Rectal Adenocarcinoma
Acronym: GCC 1314
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, PI left instituion
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00060641
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Rectal Adenocarcinoma
Keywords: Pelvic Radiotherapy; Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX (Other): Part I:
  FOLFOX: combination of drugs administered in a specific sequence as prescribed below.
  * Oxaliplatin: 85 mg/m2 intravenously (IV) over 2 hours
  * Leucovorin: 200 mg/m2 IV bolus over 2 hours
  * 5-FU: 400 mg/m2 IV bolus over 5-15 minutes, then 2,400 mg/m2 continuous IV infusion over 46-48 hours
  Part II:
  Low dose fractionated radiation therapy (LDFRT) Intensity-modulated, bone marrow sparing, whole pelvic radiation therapy 40 cGy fractions twice per day delivered at least 4-6 hours apart on the first 2 days of each chemotherapy cycle for a total of 6 cycles
  Interventions: Drug: FOLFOX {5-fluorouracil (5-FU), leucovorin, and oxaliplatin}; Radiation: Low dose fractionated radiation therapy (LDFRT)

INTERVENTIONS:
Drug: FOLFOX {5-fluorouracil (5-FU), leucovorin, and oxaliplatin} — see arm description
Radiation: Low dose fractionated radiation therapy (LDFRT) — see arm description

SUMMARY:
The purpose of this study is to assess the effects, both good and bad, of adding very low dose fractionated radiation therapy (LDFRT) to the pelvis, with FOLFOX chemotherapy prior to surgery. Standard pelvic radiation therapy given once a day (Monday through Friday) over approximately 5.5 weeks is not given in this study. You will receive 6 cycles of FOLFOX (each cycle is 2 weeks) and you will also get an LDFRT to your pelvis given twice a day on the first two days of each cycle.

DETAILED DESCRIPTION:
The current standard of care for treatment of locally advanced rectal cancer consists of neoadjuvant whole pelvic RT with radiosensitizing single-agent 5-FU followed by surgery and adjuvant full dose chemotherapy (typically FOLFOX). For all clinical T3, T4, and/or lymph node positive rectal cancer patients the standard neoadjuvant radiation dose per fraction is 180 cGy delivered on consecutive weekdays over 5.5 weeks for a total of 5040 cGy. A potentially paradigm-changing approach is currently being investigated in a phase II/III trial in which neoadjuvant RT is omitting in favor of using full dose FOLFOX chemotherapy based on provocative data published from Memorial Sloan Kettering Cancer Center. We hypothesize that whole pelvic LDFRT using 40 cGy fractions for a total of 960 cGy can be safely added concurrently to neoadjuvant full dose FOLFOX as an alternative to standard neoadjuvant 5-FU chemoradiation. We further hypothesize that using LDFRT as a chemopotentiatior will significantly increase the pCR rate as reported by the Memorial Sloan Kettering pilot study of 27%. Lastly, due to the significantly lower radiation dose per fraction and lower total radiation dose we expect that this novel strategy will not cause higher rates of severe toxicity compared to neoadjuvant FOLFOX alone.

Specifically, this phase II trial intends to determine whether 6 cycles of neoadjuvant FOLFOX with concurrent LDFRT followed by comprehensive restaging and TME achieves favorable outcomes for patients with T3N0M0, T3N1M0, or T2N1M0 rectal cancer. As mentioned above, the current standard of care for all locally advanced rectal cancer patients includes radiosensitizing 5-FU and concurrent whole pelvic RT to 5040 Gy in 180 Gy once daily fractions. Per the proposed protocol, T3N0M0, T3N1M0, or T2N1M0 rectal cancer patients who are eligible to undergo a low anterior resection would receive whole pelvic RT to 960 cGy in 40 cGy fractions delivered twice daily on days 1-2 of each cycle of FOLFOX chemotherapy for a total of 6 cycles.

Eligible study subjects include adults who are candidates for curative intent sphincter-sparing surgery and who lack high-risk features, particularly tumor encroaching upon the mesorectal fascia (within 3 mm) as determined by pre-treatment endoscopic ultrasound (EUS) and/or magnetic resonance imaging (MRI) or distal rectal tumors (<5 cm from the anal verge).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at diagnosis.
2. ECOG Performance Status 0, 1, or 2.
3. Biopsy-proven diagnosis of rectal adenocarcinoma.
4. Radiographically measurable or clinically evaluable disease by CT scan of chest/abdomen/pelvis with and without contrast ≤ 28 days prior to registration.
5. Clinical AJCC 7th edition stage T2N1M0, T3N0M0 or T3N1M0 based on physical examination, CT scan chest/abdomen/pelvis, and pelvic MRI or endorectal ultrasound.
6. Preoperative proctoscopy confirming tumor extent as no less than 5 cm and no greater than 12 cm from the anal verge.
7. Evaluation by a surgical oncologist, radiation oncologist, and medical oncologist ≤ 28 days prior to registration.
8. Confirmation by a surgeon that the patient is able to undergo a low anterior resection with total mesorectal excision ≤ 28 days prior to registration.
9. In the absence of a being treated on a clinical trial, the patient would be recommended to receive neoadjuvant chemoradiation followed by curative intent surgery.
10. The following laboratory values obtained ≤ 28 days prior to registration:

    * Absolute neutrophil count (ANC) ≥ 1500/mm3.
    * Platelet count ≥ 100,000/mm3.
    * Hemoglobin > 8.0 g/dL. May transfuse to meet eligibility.
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
    * SGOT (AST) ≤ 3 x ULN.
    * SGPT (ALT) ≤ 3 x ULN.
    * Creatinine ≤ 1.5 x ULN.
11. Negative pregnancy test (B-HCG) within 7 days prior to registration for women of childbearing potential.
12. Did the patient provide study-specific informed consent prior to study entry?
13. Willingness to return to the enrolling medical site for all study assessments.

Exclusion Criteria:

1. Clinical T4 tumor.
2. Primary surgeon indicates the need for an abdominal perineal resection (APR) at baseline.
3. Previous pelvic RT.
4. Autoimmune disease such as scleroderma, lupus, or inflammatory bowel disease.
5. Tumor < 3 mm from the mesorectal fascia as seen on MRI or endorectal ultrasound.
6. Tumor-induced symptomatic bowel obstruction.
7. Chemotherapy (including hormonal therapy) within the past 5 years from date of registration.
8. Other invasive malignancies within past 5 years from date of registration.
9. Pregnant or nursing women.
10. Men or women of childbearing potential who are unwilling to employ adequate contraception.
11. Other co-morbid conditions that, based on the judgment of the physicians obtaining informed consent, would make the patient inappropriate for this study.
12. Any conditions that would preclude a patient from completing all study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahed Badiyan, MD, Principal Investigator — UMMC MSGCC
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX: Part I:
  FOLFOX: combination of drugs administered in a specific sequence as prescribed below.
  * Oxaliplatin: 85 mg/m2 intravenously (IV) over 2 hours
  * Leucovorin: 200 mg/m2 IV bolus over 2 hours
  * 5-FU: 400 mg/m2 IV bolus over 5-15 minutes, then 2,400 mg/m2 continuous IV infusion over 46-48 hours
  Part II:
  Low dose fractionated radiation therapy (LDFRT) Intensity-modulated, bone marrow sparing, whole pelvic radiation therapy 40 cGy fractions twice per day delivered at least 4-6 hours apart on the first 2 days of each chemotherapy cycle for a total of 6 cycles
  FOLFOX {5-fluorouracil (5-FU), leucovorin, and oxaliplatin}: see arm description
  Low dose fractionated radiation therapy (LDFRT): see arm description
Period: Overall Study
Arm/Group | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 64 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure (Overall Survival Rate)
Description: Overall survival rate of patients who receive a neoadjuvant full dose FOLFOX plus the addition of concurrent LDFRT result in a pCR response rate of at least 35%.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Secondary Outcome Measure (Number of Adverse Events)
Description: Number of adverse events caused from the administration of neoadjuvant concurrent LDFRT-FOLFOX while maintaining a high rate of pelvic R0 resection compared to standard preoperative chemoradiation and total mesorectal excision surgery.
Time Frame: 1 year
Measure: Number; unit: Adverse Events
Arm/Group | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX
Number analyzed (Participants) | 3
Adverse Events | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were completing active treatment (approximately 6 weeks) and post-treatment (up to 13 additional weeks).
Arm/Group | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX (N=3)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1
White Blood Cell Decreased (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pelvic Radiotherapy With Concurrent Neoadjuvant FOLFOX (N=3)
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Platelet count Decreased (Blood and lymphatic system disorders) | 3
White Blood Cell Decreased (Blood and lymphatic system disorders) | 3
Fever (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02319304/Prot_SAP_000.pdf